CLINICAL TRIAL: NCT02057770
Title: A Pilot Study of Myeloablative Allogeneic or Haploidentical Stem Cell Transplantation With High Dose PT-Cy in Relapsed/Refractory AML
Brief Title: Allogeneic or Haploidentical Stem Cell Transplant Followed By High-Dose Cyclophosphamide in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201401080
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; fludarabine phosphate; FAMP protocol; Whole-Body Irradiation; Stem Cell Transplantation; Cyclophosphamide; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (preparative regimen, transplant, cyclophosphamide) (Experimental): BUSULFAN AND FLUDARABINE BASED PREPARATIVE REGIMEN: Patients receive busulfan IV over 3 hours on days -7 to -4, fludarabine phosphate IV over 30-60 minutes on days -6 to -2, and cyclophosphamide IV over 60 minutes on days -3 and -2.
  OR
  FLUDARABINE AND TBI BASED PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30-60 minutes on days -6 to -4 and undergo TBI twice daily on days -3 to 0.
  AND
  DONOR CELL INFUSION: Patients undergo HLA-matched sibling stem cell transplant, HLA-matched unrelated, or HLA-haploidentical transplant on day 0.
  AND
  POST-TRANSPLANT CYCLOPHOSPHAMIDE: Patients receive cyclophosphamide IV over 90 minutes on days 3 and 4.
  Interventions: Drug: busulfan; Drug: fludarabine phosphate; Radiation: total-body irradiation (TBI); Procedure: Stem cell transplant; Drug: cyclophosphamide
- CRS preventive regimen (Experimental): The final ~15 people enrolled who will be recipients of haploidentical transplants will receive tocilizumab IV over 60 minutes 6-12 hours prior to the start of the donor cell infusion.
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: busulfan
  Other Names: Myleran®
  Arms: Treatment (preparative regimen, transplant, cyclophosphamide)
Drug: fludarabine phosphate
  Other Names: Fludara®; 2-Fluoro-ara-A Monophosphate; 2-Fluoro-ara AMP, FAMP
  Arms: Treatment (preparative regimen, transplant, cyclophosphamide)
Radiation: total-body irradiation (TBI)
  Arms: Treatment (preparative regimen, transplant, cyclophosphamide)
Procedure: Stem cell transplant
  Arms: Treatment (preparative regimen, transplant, cyclophosphamide)
Drug: cyclophosphamide
  Other Names: Cytoxan®; CPM; CTX; CYT
  Arms: Treatment (preparative regimen, transplant, cyclophosphamide)
Drug: tocilizumab
  Other Names: anti-IL-6 monoclonal antibody; Actemra
  Arms: CRS preventive regimen

SUMMARY:
The purpose of this research study is to look at overall health status and how acute myeloid leukemia (AML) responds to a stem cell transplant when followed with cyclophosphamide. Some participants enrolling in this study may receive a transplant from a sibling, some may receive a transplant from a matched unrelated donor, and some may receive what is called a haploidentical transplant. A haploidentical stem cell transplant is a type of transplant that occurs when a person who needs a transplant cannot find a donor who exactly matches their tissue type (either among family members or through a matched unrelated donor). When no matched donor is available, half-matched related (haploidentical) donors may be used. Haploidentical donors are first degree relatives such as siblings, children, or parents.

People who undergo a stem cell transplant can experience complications such as rejection of the stem cell transplant or severe graft-versus-host disease (GVHD). GVHD occurs when some of the cells from the donor attack the recipient's tissues, resulting in mild, moderate, or even life-threatening side effects to the recipient's skin, stomach, intestines, and liver. However, recent research has shown that receiving cyclophosphamide after stem cell transplant can improve the outcomes of the transplant, and that is the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* AML without complete remission (CR/CRc/CRi) after at least 2 induction therapies OR
* AML that has relapsed within 6 months after obtaining a CR OR
* AML that has relapsed more than 6 months after obtaining a CR, and has treatment failure (TF) or progressive disease (PD) following at least 1 re-induction regimen OR
* AML that has relapsed post Allogeneic transplantation
* Active AML (bone marrow blasts ≥ 5% by morphology, staining, or flow) and/or presence of estramedullary disease
* Available HLA-haploidentical donor that meets the following criteria:

  * Blood-related family member (sibling (full or half), offspring, or parent, cousin, niece or nephew, aunt or uncle, or grandparent)
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by at least low-resolution typing per institutional standards
  * In the investigator's opinion, is in general good health, and medically able to tolerate leukapheresis required for harvesting HSC
  * No active hepatitis
  * Negative for HTLV and HIV
  * Not pregnant

NOTE: there were HLA-matched sibling and HLA-matched unrelated donor cohorts, but those closed without completion of accrual with Amendment 11

* Karnofsky performance status ≥ 50 %
* Adequate organ function as defined below:

  * Total bilirubin ≤ 2.5 mg/dl (unless the patient has a history of Gilbert's syndrome)
  * AST(SGOT) and ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ 2.0 x IULN OR estimated creatinine clearance ≥ 30 mL/min/1.73 m2 by Cockcroft-Gault Formula
  * Oxygen saturation ≥ 90% on room air
  * LVEF ≥ 40%
  * FEV1 and FVC ≥ 40% predicted, DLCOc ≥ 40% predicted. If DLCO is < 40%, patients will still be considered eligible if deemed safe after a pulmonary evaluation.
* At least 18 years of age at the time of study registration
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* Circulating blast count ≥ 10,000/uL by morphology or flow cytometry (cytoreductive therapies including leukapheresis or hydroxyurea are allowed)
* Known HIV or Active hepatitis B or C infection
* Known hypersensitivity to one or more of the study agents
* Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug (Day -7)
* Currently receiving or has received any intensive chemotherapy within the 14 days prior to the first dose of study drug (Day -7) (hydrea or other non-intensive regimens such as decitabine may be used but must stop at least one day prior to the first dose of study drug)
* Pregnant and/or breastfeeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) rate | Assessed at 100 days post-transplant
  The time from date of first dose of the preparative regimen until failure to engraft, treatment failure, disease progression/relapse, or death from any cause (whichever occurs first). Rates will be calculated with exact 95% confidence intervals.

SECONDARY OUTCOMES:
Overall Survival (OS) | Assessed at 1 year post-transplant
  The time from the date of day 0 until death from any cause. Rates will be calculated with exact 95% confidence intervals.
Rate of Leukemia Free Survival (LFS) | Assessed at 100 days post-transplant
  The time from date of day 0 until disease progression or death from any cause (whichever occurs first). Rates will be calculated with exact 95% confidence intervals. For patients who achieve CR, CRc, or CRi only.
Transplant Related Mortality (TRM) Rate | Assessed at 100 days post-transplant
  Death from causes other than disease relapse or progression prior to Day +100 visit. Rates will be calculated with exact 95% confidence intervals.
Time to neutrophil engraftment | Assessed up to day 30
  Defined as an untransfused platelet measurement > 20,000/ x10^9/L x 3 consecutive days. Kaplan-Meier models will be used to estimate median time to platelet engraftment and plot a time to event curve. Cox proportional hazards models may be used to explore the effect of covariates on time to platelet engraftment.
Incidence of acute GVHD | Up to 100 days post-transplant
  The incidence and severity of acute GVHD will be determined. Rates will be calculated with exact 95% confidence intervals.
Incidence of chronic GVHD | 1 year post-transplant starting at day +100
  The incidence and severity of chronic GVHD will be determined. Rates will be calculated with exact 95% confidence intervals.
Time to platelet engraftment | Assessed up to day 100
  Defined as an untransfused platelet measurement > 20,000/ x10^9/L x 3 consecutive days. Kaplan-Meier models will be used to estimate median time to platelet engraftment and plot a time to event curve. Cox proportional hazards models may be used to explore the effect of covariates on time to platelet engraftment.
Rate of CRS with and without tocilizumab prophylaxis | Assessed up to day 7
  To investigate the rate of cytokine release syndrome with and without tocilizumab prophylaxis in patients with active AML who undergo haploidentical transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Todd Fehniger, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu